CLINICAL TRIAL: NCT06311929
Title: VETC-based Precision Adjuvant Therapy for Postoperative Hepatocellular Carcinoma: a Prospective Multicenter Cohort Study
Brief Title: Precision Adjuvant Therapy After Surgery for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Precision AT-01
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: HCC
Keywords: HCC; Adjuvant therapy; VETC; PD-1 inhibitor; Lenvatinib
MeSH Terms: interventions — lenvatinib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined adjuvant therapy group (Experimental): Patients in the combined adjuvant therapy group received PD-1 monoclonal antibody with Lenvatinb adjuvant therapy after liver resection.
  Interventions: Drug: PD-1 monoclonal antibody and lenvatinib
- Monotherapy group (Active Comparator): Patients in the monotherapy group received PD-1 monotherapy after liver resection.
  Interventions: Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: PD-1 monoclonal antibody and lenvatinib — Patient receives first adjuvant PD-1 monoclonal antibody 2-4 weeks postoperatively, 200 mg IV, every 21 days for a total of 9 cycles; lenvatinib is initiated orally 2-4 weeks postoperatively for 6 months.
  Other Names: Non
  Arms: Combined adjuvant therapy group
Drug: PD-1 monoclonal antibody — Patient receives first adjuvant PD-1 monoclonal antibody 2-4 weeks postoperatively, 200mg IV over 21 days for 9 cycles.
  Other Names: Non
  Arms: Monotherapy group

SUMMARY:
Vessels that encapsulate tumor clusters (VETC) is an invasive metastatic factor in HCC independent of the epithelial mesenchyme transition (EMT), and VETC-positive patients have a higher rate of postoperative recurrence. How to improve the prognosis of this group of patients is an urgent issue to be addressed.

DETAILED DESCRIPTION:
Previous studies have identified VETC as a new metastatic pattern independent of EMT that may be associated with immunosuppression as well as poor prognosis. Multiple retrospective studies find higher rates of postoperative recurrence, distant metastasis in VETC-positive patients. How to improve surgical prognosis in VETC-positive patients needs to be explored. There are no published studies on how to improve prognosis for this population. One of our unpublished retrospective studies found that VETC-positive patients receiving PD-1 monoclonal antibody was not effective in improving prognosis. However, PD-1 monoclonal antibody in combination with PD-1 monoclonal antibody effectively reduced postoperative recurrence and improved prognosis in VETC-positive patients. Based on our previous retrospective data, this multicenter prospective cohort study was designed to further validate and explore effective therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75.
2. No previous local or systemic treatment for hepatocellular carcinoma.
3. Child-Pugh liver function score ≤ 7.
4. ECOG PS 0-1.
5. No serious organic diseases of the heart, lungs, brain, kidneys, etc.
6. Pathologic type is hepatocellular carcinoma.
7. Confirmation of the presence of VETC vascular pattern by CD34 immunohistochemical staining.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Suffering from a condition that interferes with the absorption, distribution, metabolism, or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, impaired absorption, etc.).
3. A history of gastrointestinal bleeding within the previous 4 weeks or a definite predisposition to gastrointestinal bleeding (e.g., known locally active ulcer lesions, fecal occult blood ++ or more, or gastroscopy if persistent fecal occult blood +) that has not been targeted, or other conditions that may have caused gastrointestinal bleeding (e.g., severe fundoplication/esophageal varices), as determined by the investigator.
4. Active infection.
5. Other significant clinical and laboratory abnormalities that affect the safety evaluation.
6. Inability to follow the study protocol for treatment or follow up as scheduled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of include in this research until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  DFS defined as time to recurrence or death after surgery.

SECONDARY OUTCOMES:
Overall survival | From date of include in this research until the date of death from any cause, whichever came first, assessed up to 60 months
  OS defined as time to death from any cause after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code